CLINICAL TRIAL: NCT04409132
Title: A Randomized 4 Period Study to Investigate the Pharmacokinetic Comparability of Dosing Triferic AVNU IV by Continuous Infusion and IV Bolus.
Brief Title: Study to Investigate the Pharmacokinetic Comparability of Dosing Triferic AVNU IV by Continuous Infusion and IV Bolus.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-26
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-04

CONDITIONS: End Stage Renal Disease
Keywords: Pharmacokinetics
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Triferic AVNU infusion pre-dialyzer (Experimental): Patients will receive one (1) 6.75 mg Fe dose of Triferic AVNU by continuous infusion over 3 hours into the predialyzer blood line.
  Interventions: Drug: Triferic
- Triferic AVNU for injection at T=0 and T= 3 hours (Experimental): Patients will receive two (2) doses of Triferic AVNU 3.4 mg IV (2.25 mL) at T=0 and T=3 hours of hemodialysis into the venous drip chamber.
  Interventions: Drug: Triferic
- Triferic AVNU for injection at T=0 (Experimental): Patients will receive one (1) dose of Triferic AVNU 0.08 mg/kg IV, up to 6.75 mg Fe, at T=0 of hemodialysis into the venous drip chamber.
  Interventions: Drug: Triferic
- Triferic AVNU for injection at T=0, T=1.5 and T= 3 hours (Experimental): Patients will receive three (3) doses of Triferic AVNU 2.25 mg Fe (1.5 mL) at T=0, T=1.5 and T=3.0 hours of hemodialysis into the venous drip chamber.
  Interventions: Drug: Triferic

INTERVENTIONS:
Drug: Triferic — Triferic (ferric pyrophosphate citrate, FPC), an iron-replacement product, is an iron complex in which iron(III) is bound to pyrophosphate and citrate.
  Other Names: ferric pyrophosphate citrate; FPC

SUMMARY:
This study will investigate the administration of Triferic AVNU intravenously by three different administration schedules compared to continuous infusion over 3 hours

DETAILED DESCRIPTION:
An open-label, randomized, four period sequential study of Triferic AVNU administered intravenously by three different administration schedules compared to continuous infusion over 3 hours

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients ≥18 years of age.
* Signed informed consent to participate in the study.
* Stable on hemodialysis prescription for ≥3 months.
* Able to sustain hemodialysis 3x/week for 3 to 4 hours.
* Hemoglobin concentration >9.5 g/dL.
* Serum TSAT ≥20%.
* Receiving hemodialysis via AV fistula or graft.
* Able to receive hemodialysis for 4 hours at each session over the duration of the treatment periods.
* Able to receive intermittent heparin administration for anticoagulation of the dialysis circuit.
* Serum TIBC ≥ 150 µg/dL.

Exclusion Criteria:

* Active bleeding disorder (GI, skin, nasal…)
* Receiving hemodialysis via catheter.
* Receiving IV iron within 10 days of the first on-study hemodialysis treatment.
* Receiving oral iron within 10 days of the first on-study hemodialysis treatment.
* Any other condition, that in the opinion of the investigator would not allow completion of the 4 hemodialysis treatments in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve (AUC0-last pFetotal) for all Treatments A,B,C and D | 8 hours
Area under plasma transferrin bound plasma iron concentration- time curve (AUC0-last FeTBI) for all Treatments A,B,C and D | 8 hours

SECONDARY OUTCOMES:
Maximum observed plasma iron concentration (Cmax pFetotal) for all Treatments A,B,C and D | 8 hours
Maximum observed transferrin bound plasma iron concentration (Cmax FeTBI) for all Treatments A,B,C and D | 8 hours
Maximum observed serum iron concentration (Cmax sFetotal) for all Treatments A,B,C and D | 8 hours
Area under serum Fe concentration-time curve (AUC0-last sFetotal) for all Treatments A,B,C and D | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No